CLINICAL TRIAL: NCT06909474
Title: Clinical Study of CD5 Targeting Chimeric Antigen Receptor NK Cells (CAR-NK) in the Treatment of Relapse/Refractory T-Cell Hematologic Malignancies
Brief Title: Clinical Trial of CD5-targeted CAR-NK Therapy for Relapse/Refractory T-Cell Hematologic Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chongqing Precision Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBC083
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: T-ALL/Lymphoma
Keywords: T-ALL; T-LBL; PTCL-NOS; AITL; ALCL; ENKL; T-PLL; ATLL; MF/SS
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia-Lymphoma, Adult T-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CD5 CAR-NK cells (Experimental)
  Interventions: Biological: Anti-CD5 CAR NK cells

INTERVENTIONS:
Biological: Anti-CD5 CAR NK cells — Each patient will initially receive a single infusion of CAR-NK cells on Day 0. If a suboptimal response is observed after the first infusion (assessed by Day 28) and the safety profile remains acceptable, a second infusion may be administered as a remedial dose after Day 28. CAR-NK cells need to be controlled within 70 minutes from thawing to infusion completion.

SUMMARY:
This is a clincal trial initiated by investigator to evaluate the safety and efficacy of anti-CD5 CAR-NK in the treatment of patients with relapsed/refractory T-Cell hematologic malignancies.

DETAILED DESCRIPTION:
This study is a single-arm, open-label, dose-finding and expansion clinical trial aimed at evaluating the safety and efficacy of anti-CD5 CAR-NK therapy for the treatment of patients with relapsed/refractory T-Cell hematologic malignancies. The goal is to determine the recommended dose of CAR-NK cell therapy for these conditions. The study includes three dose groups: 1×10⁷ CAR-positive cells/kg, 3×10⁷ CAR-positive cells/kg, and 5×10⁷ CAR-positive cells/kg. Each patient will initially receive a single infusion of CAR-NK cells on Day 0. If a suboptimal response is observed after the first infusion (assessed by Day 28) and the safety profile remains acceptable, a second infusion may be administered as a remedial dose after Day 28. The investigaors have the flexibility to adjust the second infusion dose based on the subject's condition.

ELIGIBILITY:
Inclusion Criteria:

-

1.Gender and Age: No gender restriction; age 18-75 years (inclusive). 2.Diagnosis: Confirmed diagnosis of T-cell acute lymphoblastic leukemia (T-ALL) or T-cell lymphoma, including:

1. T-ALL Patients: Bone marrow morphology during screening shows ≥5% blasts/immature lymphocytes and/or flow cytometry confirms minimal residual disease (MRD)+, and meets any of the following:

   1. Refractory to ≥2 cycles of standard induction chemotherapy (failure to achieve CR).
   2. Relapsed within 12 months after achieving CR with first-line induction therapy.
   3. Failure to achieve CR or relapse after ≥2 lines of chemotherapy.
   4. Relapse after hematopoietic stem cell transplantation (HSCT).
2. T-cell Lymphoma Patients: Confirmed diagnosis of T-lymphoblastic lymphoma (T-LBL) or T-cell non-Hodgkin lymphoma (including but not limited to: peripheral T-cell lymphoma, not otherwise specified (PTCL-NOS), angioimmunoblastic T-cell lymphoma (AITL), anaplastic large cell lymphoma (ALCL), extranodal NK/T-cell lymphoma (ENKL), T-cell prolymphocytic leukemia (T-PLL), adult T-cell leukemia/lymphoma (ATLL), mycosis fungoides/Sézary syndrome (MF/SS) stage IIB or higher), and meets both:

   1. At least one bidimensionally measurable lesion per Lugano 2014 criteria: nodal lesions >1.5 cm in long axis; extranodal lesions >1.0 cm in long axis.
   2. Refractory to ≥2 lines of chemotherapy, primary resistance, or relapse post-HSCT.

      3.CD5 Positivity: Confirmed by flow cytometry (≥80% tumor cells express CD5 with mean fluorescence intensity [MFI] equivalent to normal T cells; Dim defined as MFI ≥1 log lower than normal T cells; partial positivity defined as 20-80% tumor cells expressing CD5) or immunohistochemistry (>30% tumor cells express CD5).

      4.ECOG Performance Status: 0-2 . 5.Life Expectancy: ≥12 weeks. 6.Organ Function:

   <!-- -->

   1. Cardiac: Left ventricular ejection fraction (LVEF) ≥50% by echocardiography; no significant ECG abnormalities.
   2. Renal: Serum creatinine ≤2.0×ULN.
   3. Hepatic: ALT/AST ≤3.0×ULN (≤5.0×ULN if liver involvement); total bilirubin ≤2.0×ULN.
   4. Pulmonary: Oxygen saturation ≥92% (room air). 7.No Contraindications: To leukapheresis, venipuncture, or cell collection. 8.No Severe Psychiatric Disorders. 9.Contraception: Agreement to use effective contraception from informed consent until 1 year post-CAR-NK infusion (for patients of childbearing potential).

      10.Informed Consent: Signed by the patient or legal guardian, confirming understanding of the trial's purpose and procedures.

Exclusion Criteria:

1. Prior CAR-NK therapy or genetically modified cell therapy.
2. Active CNS involvement at screening (prior CNS involvement with resolved status post-treatment is allowed).
3. Recent Anticancer Therapy:

   1. Chemotherapy, targeted therapy, or investigational drugs within 2 weeks or 5 half-lives prior to screening.
   2. Radiotherapy within 2 weeks prior to screening.
4. Active/Uncontrolled Infection: Within 1 week prior to screening.
5. Cerebrovascular Event or Seizure: Within 6 months prior to screening.
6. Viral Infections:

   1. HBV DNA > ULN (if HBsAg+ or HBcAb+).
   2. HCV RNA > ULN (if HCV Ab+).
   3. HIV+, syphilis+, or active tuberculosis.
7. Cardiac Disease:

   1. NYHA Class III/IV congestive heart failure.
   2. Myocardial infarction or CABG ≤6 months prior.
   3. Clinically significant ventricular arrhythmia or unexplained syncope (excluding vasovagal/dehydration-related).
   4. Severe cardiomyopathy.
8. Active/Uncontrolled Autoimmune Disease.
9. Prior Malignancy: Within 5 years, except for cured cervical carcinoma in situ, basal/squamous skin cancer, localized prostate cancer, or ductal carcinoma in situ.
10. Live Vaccination: Within 4 weeks prior to screening.
11. Pregnancy/Lactation: Pregnant, breastfeeding, or planning pregnancy within 1 year post-CAR-NK infusion.
12. Other: Investigator-determined ineligibility.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 28 dyas
  The incidence of adverse events after CAR-NK cell infusion was assessed by CTCAE, version 5.0.
Objective response rate (ORR) | 1month, 2 months, 3 months
  Objective Response Rate (ORR) within 3 Months:
  1. For patients with T-cell lymphoma, ORR includes complete response (CR) and partial response (PR);
  2. For patients with T-cell acute lymphoblastic leukemia (T-ALL), ORR includes CR, CR with partial hematologic recovery (CRh), CR with incomplete hematologic recovery (CRi), and morphologic leukemia-free state (MLFS).
Overall survival (OS) after CAR-NK infusion | 2 years
  OS is defined as the time from CAR-NK cell infusion to death from any cause, reflecting the long-term survival benefit of the therapy.
Duration of response (DOR) after CAR-NK infusion | 2 years
  DOR measures the time from the first achievement of objective response to disease progression or death, evaluating the durability of treatment efficacy in responding patients.
Progression-Free-Survival (PFS) after CAR-NK infusion | 2 years
  PFS is the time from CAR-NK cell infusion to disease progression or death from any cause, capturing both tumor control and survival outcomes

SECONDARY OUTCOMES:
To obtain the cytodynamics data of CAR-NK cells in vivo【pharmacokinetics】 | 3months
  Cmax:The highest concentration of CAR T cells amplified in peripheral blood after reinfusion
To obtain the cytodynamics data of CAR-NK cells in vivo【pharmacokinetics】 | 3months
  Tmax:The time to reach the highest concentration of CAR-NK cells in peripheral blood after reinfusion
To obtain the cytodynamics data of CAR-NK cells in vivo【pharmacodynamics】 | 3months
  The content of free IL-6 in peripheral blood at each time point after transfusion was determined by immunohistochemical method

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei, China